CLINICAL TRIAL: NCT01237405
Title: Study of 99mTc-EC20 Imaging (FolateScan) in Participants With Knee Osteoarthritis
Brief Title: A Study of FolateScan in Patients With Knee Osteoarthritis
Status: Completed | Type: Observational
Sponsor: Virginia Kraus (Other)
Collaborators: Eli Lilly and Company (Industry); Endocyte (Industry)
Responsible Party: Sponsor-Investigator, Virginia Kraus, Professor, Duke University
Organization: Duke University (Other)
Other Study IDs: Pro00018123; Protocol H7L-MC-MDAB(b) (Other Grant/Funding Number: Eli Lilly and Company)
Record Dates: First submitted 2010-10-26; First posted 2010-11-09 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthritis; nuclear medicine; macrophages
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, serum, urine, synovial fluid
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Knee Osteoarthritis: Unilateral or bilateral knee osteoarthritis on radiograph associated with knee pain on most days of any one-month in the last year in at least one knee.
  Study participants underwent a one-time evaluation by FolateScan which entailed a single intravenous injection of 99mTc-EC20 (total volume of 1.0 to 2.0 ml administered over a period of 30 seconds with radioactive dose between 20 and 25 mCi).
  Interventions: Drug: 99mTc-EC20

INTERVENTIONS:
Drug: 99mTc-EC20 — Study participants underwent a one-time evaluation by FolateScan which entailed a single intravenous injection of 99mTc-EC20 (total volume of 1.0 to 2.0 ml administered over a period of 30 seconds with radioactive dose between 20 and 25 mCi). A total of three imaging scans were acquired: an early phase (at ~1 minute) SPECT/CT of both knees; a late phase (at ~60 minutes) SPECT/CT image of both knees; and a late phase (at ~80 minutes) planar image of the whole body was performed (anterior-posterior, and postero-anterior).
  Other Names: (FolateScan Imaging Drug)

SUMMARY:
The purpose of this study is to evaluate 99mTc - EC20 imaging (FolateScan), a Nuclear Medicine imaging technology that enables localization of activated macrophages in the joints of participants with knee osteoarthritis (OA). Twenty five participants with symptomatic unilateral or bilateral knee OA will undergo a one-time evaluation of the knee as follows: knee radiography, FolateScan of the knees and whole body, musculoskeletal exam, questionnaires, sampling of blood, urine and synovial fluid for analysis of inflammatory markers. Data analysis will be cross-sectional and include a comparison of the location and intensity of EC20 uptake with the following: radiographic knee OA severity, clinical measures of disease severity, cytokine expression, and synovial fluid cell count.

DETAILED DESCRIPTION:
Each study day will on average last one day per individual and each individual will be followed for development of an Adverse Event for 7 days

ELIGIBILITY:
Inclusion Criteria: Unilateral or bilateral knee OA; Kellgren Lawrence grade 1-4; Knee pain on most days of any one-month in the last year in at least one knee; Age > 18 years old.

Exclusion Criteria: Arthroscopic knee surgery within the previous 12 months; Intra-articular injection or systemic (oral, IV, IM) steroid within previous 6 months; Any knee replacement; Current enrollment in, or discontinued within the last 30 days from, a clinical trial involving an off-label use of an investigational drug or device (other than the study drug used in this study); Pregnancy; Positive serum beta HCG within 48 hours prior to 99mTc-EC20 administration and/or lactation; Rheumatoid arthritis or other inflammatory arthropathy; Avascular necrosis; Periarticular fracture; Current anticoagulant therapy; Current immune modulator therapy, or any such therapy within 4 weeks of study procedures; Inability to discontinue use of NSAIDS within 3 days of study procedures (low dose aspirin of up to 325 mg per day is permitted); Must be able to stop Folic Acid containing vitamins 24 hrs before study; Paget's disease; Villonodular synovitis; Joint infection; Ochronosis; Neuropathic arthropathy; Acromegaly; Hemochromatosis; Wilson's disease; Osteochondromatosis; Personnel directly affiliated with this study or their immediate family members; Concurrently enrolled in any other type of medical research judged not to be scientifically or medically compatible with this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Males and females over the age of 18 years with at least one symptomatic knee with evidence of osteoarthritis on radiograph.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2010-10; Primary Completion 2011-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Frequency of knee uptake of 99mTc-EC20 | Baseline
  These data will be collected at a single timepoint (baseline) only and participants will not be further followed.

SECONDARY OUTCOMES:
Intensity and location of uptake of 99mTc-EC20 | Baseline
  These data will be collected at a single timepoint (baseline) only and participants will not be further followed.
Correlation of knee symptoms and knee uptake of 99mTc-EC20 | Baseline
  This analysis will be performed from data collected at a single timepoint (baseline) only and participants will not be further followed.
Correlation of 99mTc-EC20 uptake and biomarkers | Baseline
  This analysis will be performed from data collected at a single timepoint (baseline) only and participants will not be further followed.
Correlation of knee radiographic OA and knee uptake of 99mTc-EC20 | Baseline
  This analysis will be performed from data collected at a single timepoint (baseline) only and participants will not be further followed.

CONTACTS AND LOCATIONS:
Overall Officials: Virginia B Kraus, MD, PhD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

REFERENCES:
- [Result] Matteson EL, Lowe VJ, Prendergast FG, Crowson CS, Moder KG, Morgenstern DE, Messmann RA, Low PS. Assessment of disease activity in rheumatoid arthritis using a novel folate targeted radiopharmaceutical Folatescan. Clin Exp Rheumatol. 2009 Mar-Apr;27(2):253-9. PMID 19473565
- [Derived] Haraden CA, Huebner JL, Hsueh MF, Li YJ, Kraus VB. Synovial fluid biomarkers associated with osteoarthritis severity reflect macrophage and neutrophil related inflammation. Arthritis Res Ther. 2019 Jun 13;21(1):146. doi: 10.1186/s13075-019-1923-x. PMID 31196179
- [Derived] Kraus VB, McDaniel G, Huebner JL, Stabler TV, Pieper CF, Shipes SW, Petry NA, Low PS, Shen J, McNearney TA, Mitchell P. Direct in vivo evidence of activated macrophages in human osteoarthritis. Osteoarthritis Cartilage. 2016 Sep;24(9):1613-21. doi: 10.1016/j.joca.2016.04.010. Epub 2016 Apr 12. PMID 27084348